CLINICAL TRIAL: NCT01037296
Title: Catheter Ablation of Atrial Fibrillation Using Hansen Medical Robotic Navigation - A Randomised Controlled Trial
Brief Title: Catheter Ablation of Atrial Fibrillation Using Hansen Medical Robotic Navigation
Acronym: Hansen
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Based on interim analysis study felt unlikely to reach the primary aim
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005815
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; robotic navigation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- manual ablation (Other)
  Interventions: Procedure: catheter ablation
- robotic ablation (Experimental)
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — ablation procedure performed with Hansen robotic navigation system
  Arms: robotic ablation
Procedure: catheter ablation — Ablation will be performed as normal treatment
  Arms: manual ablation

SUMMARY:
Atrial fibrillation (AF) affects as many as 1 in 100 people and reduces the quality of life of large numbers of people in the UK and around the world. Catheter ablation is a minimally invasive treatment that has been developed to help eliminate AF. It is a complex procedure to perform so only a few hospitals are able to offer this treatment in the UK. A new technology allows the operator to guide their catheters (thin wires) in the patient by using a robotically steered sheath. This allows accurate and precise navigation that may improve the accuracy and integrity of ablation. We aim to prove whether this technology can make AF ablation easier and more effective.

Substudy: Platelet reactivity and activation in AF, and the impact of curative ablation. Blood and urine samples will be taken pre- and 3 months post ablation to see if platelet reactivity and activation are affected by AF compared to established normal ranges, and whether curative ablation impacts on this.

ELIGIBILITY:
Inclusion Criteria:

* All patients with symptomatic AF planned for catheter ablation.

Exclusion Criteria:

* Age < 18 years
* Previous ablation procedure
* Expected life expectancy < 6 months
* Inability or unwillingness to sign consent
* Pregnancy
* Contraindications for the ablation procedure o Thrombus in the left atrium that fails to resolve with optimal oral anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Single procedure success rate at 12 months | 12 months

SECONDARY OUTCOMES:
Complication rates, catheter stability, procedure/fluoroscopy time (and dose), subjectively assessed operator fatigue | 0-12 months
Platelet substudy: Platelet activation post ablation compared to baseline. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Barts and the London NHS Trust, London, London, United Kingdom

REFERENCES:
- [Result] Ullah W, McLean A, Hunter RJ, Baker V, Richmond L, Cantor EJ, Dhinoja MB, Sporton S, Earley MJ, Schilling RJ. Randomized trial comparing robotic to manual ablation for atrial fibrillation. Heart Rhythm. 2014 Nov;11(11):1862-9. doi: 10.1016/j.hrthm.2014.06.026. Epub 2014 Jun 21. PMID 24960268
- [Derived] Duncan ER, Finlay M, Page SP, Hunter R, Goromonzi F, Richmond L, Baker V, Ginks M, Ezzat V, Dhinoja M, Earley MJ, Sporton S, Schilling RJ. Improved electrogram attenuation during ablation of paroxysmal atrial fibrillation with the Hansen robotic system. Pacing Clin Electrophysiol. 2012 Jun;35(6):730-8. doi: 10.1111/j.1540-8159.2012.03381.x. Epub 2012 Apr 11. PMID 22494451